CLINICAL TRIAL: NCT03585192
Title: Safety of Immediate Skin-to-Skin Contact After Vaginal Birth in Vigorous Late-Preterm Neonates - A Pilot Study
Brief Title: Safety of Immediate Skin-to-Skin Contact After Vaginal Birth in Vigorous Late-Preterm Neonates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment closed due to impending graduation from Fellowship
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Rebecca Walsh, Neonatology Fellow, MD, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-17-24
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin Group (Experimental): Pulse oximeter probe is placed on right wrist of vigorous neonate after vaginal birth. If randomized to skin group, neonate will initiate skin-to-skin contact after umbilical cord is cut and dried with warm blankets on Mother's abdomen. Length of monitoring will be for first hour of life.
  Interventions: Other: Skin Group
- Warmer Group (Active Comparator): Pulse oximeter probe is placed on right wrist of vigorous neonate after vaginal birth. If randomized to warmer group, neonate will initiate skin-to-skin contact after 20 minutes of observation under the radiant warmer. Length of monitoring will be for first hour of life.
  Interventions: Other: Warmer Group

INTERVENTIONS:
Other: Skin Group — 1. If the newborn is vigorous (crying, good respiratory effort, good tone) after vaginal delivery, newborn will be able to go directly to Mother's chest for immediate SSC
  2. A pulse oximeter will be placed on the newborn's right wrist. Saturations will be monitored on a pulse oximeter located next to the Mother's bed for the first hour of life.
  Arms: Skin Group
Other: Warmer Group — 1. Newborn will go to the radiant warmer, pulse oximeter placed on newborn's right wrist, and saturations will be monitored on the Panda Warmer.
  2. If stable per Baby RN after 20 minutes of observation, the newborn will be placed on Mother's chest for SSC. Vital signs will be monitored for the first hour of life.
  Arms: Warmer Group

SUMMARY:
Late-preterm neonates are born between 34 and 36 weeks 7 days gestational age (GA). Neonates born less than 34 weeks GA are at increased risk for morbidity and directly admitted to the Neonatal Intensive Care Unit (NICU). Skin-to-skin contact (SSC) is a standard of care in many units to aid in post-natal transitioning. Current guidelines published by the Neonatal Resuscitation Program (NRP) and American Academy of Pediatrics (AAP) recommend only "vigorous, term" neonates initiate immediate SSC. There is no published data regarding safety or guidelines relating to late-preterm neonates and immediate SSC. Therefore, the investigators hypothesize that post-natal transitioning after immediate SSC within the first hours after birth will be no worse for vigorous, singleton 35 0/7 to 36 6/7 week neonates compared to those who transition to SSC after an initial period of 20 minutes observation under the radiant warmer.

DETAILED DESCRIPTION:
Aim: Determine safety of immediate skin-to-skin in vigorous 35 0/7 to 36 6/7 week late-preterm singleton neonates after vaginal delivery compared to current practice of observation under the radiant warmer for 20 minutes.

Organization - University Hospital's Cleveland Medical Center Department of Obstetrics & Gynecology and Rainbow Babies Children's Hospital Department of Neonatology will be the only participating members.

Study Design - This is a prospective, randomized-control, and equivalence study. The cohort of subjects that will be recruited for this study will include singleton neonates born via vaginal delivery to Mothers at 35 0/7 to 36 6/7 weeks GA in UH MacDonald Women's Hospital Labor & Delivery Hospital.

Recruitment Procedures

1. Recruitment will occur at UH MacDonald Women's Hospital
2. Mothers who meet the inclusion criteria will be tracked in the EMR at time of admission to the Labor & Delivery Unit.
3. Informed consent will be obtained by members of the research team.
4. Consenting process will occur at the time of Mother's admission to the Labor & Delivery Unit.
5. Consent will be obtained in Mother's room.
6. Mother will not be consented if sedated, under distress from laboring process, or clinically unstable per Labor & Delivery Team.
7. A copy of the consent will be given to the Mother, a copy kept in a locked, secure office for research collection purposes, and a copy will be scanned into the electronic medical record (EMR).

Randomization

1. Index cards with skin or warmer written on them will be placed in opaque, sealed envelopes.
2. The envelopes will be shuffled randomly and numbered 1-120. The envelopes will be kept in chronological order. Extra envelopes containing index cards will be made if needed using the same randomized process.
3. Envelopes will be stored in the Neonatal Treatment Room adjacent to Operation Room 1 on the Labor & Delivery Unit.
4. After obtaining informed consent and if the Mother is agreeable to participate in this study, a sealed envelope will be brought to the laboring room and opened prior to delivery. No one in the delivery room will know what is written on the index card. The envelope will be opened right before delivery.
5. Skin is the intervention group (Group 1) and warmer is the control group (Group 2)
6. Information about how the newborn transitioned after birth will be collected, regardless if newborn is in the skin or warmer group. The information gathered will be analyzed to determine if there are any differences in postnatal transitioning between the two groups of newborns.

Study Methods Preparation prior to vaginal delivery (all late-preterm neonates)

1. Prepare Mother to receive newborn (bra removed & uncover breasts)
2. Place warm blanket on Mother's abdomen to receive neonate.
3. Pulse oximeter will be turned on and placed bedside to allow uninterrupted contact and positioning between Mother and neonate. Screen is to be visible to Labor & Delivery RN at all times.

Initiate immediate SSC after vaginal birth of vigorous late-preterm neonate - Group 1 (skin)

1. Newborn Nurse will assist Mother with initiating skin-to-skin contact
2. Place nude neonate supine on warm blanket on Mother's abdomen
3. Suction mouth and nose if necessary, dry, & remove wet blanket
4. Place pulse oximeter on right upper extremity, hat, diaper, and cover with warm receiving blanket
5. Assign 1 minute APGAR
6. Any change in clinical status of either Mother (based on clinical judgment by OB Physician or Midwife) or neonate (based on clinical judgment by Pediatric Team or Neonate's RN) will preclude continued SSC and warrant immediate intervention until stabilized.

   1. Interventions to stabilize neonate: repositioning on Mother's chest, ensure unobstructed airway, oral suctioning with bulb syringe if needed, reapply pulse oximeter, & remove from Mother's chest if needed.

Monitoring during postnatal transitioning

1. Place neonate in prone position on Mother's bare chest between breasts in upright position within 5 minutes of birth
2. Monitor neonate's head position and ensure nose is unobstructed
3. Cover with 2-4 layers of warm receiving blankets
4. Assign 5 minute APGAR
5. Neonate to stay on Mother's chest for uninterrupted SSC for first 60-90 minutes of life or until completion of first feed
6. Routine vital signs, including pulse oximetry, will be monitored and documented in the EMR until Mother/neonate stable for transfer to antepartum unit. Vital signs will be obtained per current UH protocol. Normal values and assessment data include:

   1. Axillary temperature 36.5-37.5 degrees Celsius
   2. Heart rate of 100 to 180 beats per minute (if not eating or crying)
   3. Regular cardiac rhythm
   4. Respiratory rate of 40-60 breaths per minute
   5. Pulse oximetry parameters per NRP guidelines.
   6. Any pulse oximetry reading < 88% at 1 hour of life will require the baby to be repositioned on Mother's chest, ensure unobstructed airway, oral suctioning with bulb syringe if needed, reapply pulse oximeter, & remove from Mother's chest if needed.
   7. Screening and management of postnatal glucose homeostasis will be instituted, as is the current policy at UH MacHouse Women's Hospital, for all late-preterm neonates until 24 hours of life.
7. Signs of tolerance of postnatal SSC:

   1. Pink or with mild acrocyanosis
   2. Respiratory effort easy, no audible grunting, or visible intercostal retractions
   3. Alert, demonstrating feeding cues, or sleeping comfortably
   4. Well-flexed posture with good tone
8. Any change in clinical status of either Mother (based on clinical judgment by OB Physician or Midwife) or neonate (based on clinical judgment by Pediatric Team or Neonate's RN) will preclude continued SSC and warrant immediate intervention until stabilized.

   1. Interventions to stabilize neonate: repositioning on Mother's chest, ensure unobstructed airway, oral suctioning with bulb syringe if needed, reapply pulse oximeter, & remove from Mother's chest if needed.

Monitoring of late-preterm neonate if randomized to Group 2 (warmer)

1. Initial period of observation (20 minutes) under the radiant warmer per current UH protocol
2. Place pulse oximeter on right upper extremity
3. SSC within 1 hour after birth for at least 1 hour and until first breastfeed attempt
4. SSC protocol to be followed as detailed in (numbers 2-7)
5. Any change in clinical status of either Mother (based on clinical judgment by OB Physician or Midwife) or neonate (based on clinical judgment by Pediatric Team or Neonate's RN) will preclude continued SSC and warrant immediate intervention until stabilized.

   1. Interventions to stabilize neonate: repositioning on Mother's chest, ensure unobstructed airway, oral suctioning with bulb syringe if needed, reapply pulse oximeter, & remove from Mother's chest if needed.

Data Collection & Storage

1. Data to be de-identified once collected from the current electronic medical record and entered into a linking log in a secure file in the RedCap Database.
2. Mother and Baby will be assigned a study number.
3. If randomized into Group 1 (skin), dyad will be identified as: Mother - MS1 and Baby - S1. Each additional dyad randomized into Group 1 will continue sequentially (i.e. MS2, MS3, & S2, S3, etc.)
4. Group 2 (warmer) will be identified as: Mother - MW1 and Baby - W1. Each additional dyad randomized into Group 2 will continue sequentially (i.e. MW2, MW3, & W2, W3, etc.)
5. A separate, secure file in RedCap Database will be created for Mother's and baby's information.
6. Maternal information to be collected: medical record number, age, race, gravida/para status, prenatal screens, medical history, medications, date of delivery, time of delivery, & planned feeding method (breast or formula).
7. Neonate information to be collected: medical record number, gestational age, sex, race, Apgar scores (1, 5, & 10 minutes), time of initial SSC, & if SSC is interrupted (time & reason). Vitals, including pulse oximetry, will be collected per UH protocol. If respiratory distress is present, initial glucose level & time, time of initial feed, and time of transfer & location (postpartum unit or NICU with admission diagnosis).
8. All of the above information will be collected throughout the entire hospital admission.
9. The investigators will also track any NICU admission and document reason for admission.
10. A data safety monitoring committee will periodically review the collected data to ensure continued safety during ongoing trial.

Statistical Analysis & Power Calculations

The investigators will test the hypothesis that Apgar scores at 1, 5 and 10 minutes, temperature at each measured time, presence of respiratory distress and oxygen saturation is not worse among the SSC babies compared to those with the standard of care (warmer).

Means and standard deviations will be calculated for continuous variables, median and ranges for scores, and counts and percentages for categorical variables. Differences between babies in the two randomization groups will be analyzed using a t-test (for continuous variables, such as temperature), a wilcoxon rank sum test (for ordinal variables, such as Apgar scores) or chi-square test for categorical variables (such as presence of respiratory distress). Prior to analysis, data will be tested for consistency with test assumptions and alternatives (such as Fisher's exact instead of chi-square) will be used if more appropriate. P-values will be one sided and a p<0.05 will be used to reject our hypothesis of non-inferiority.

Additional variables, such as characteristics of the Mother, can be analyzed in a similar fashion for exploratory analyses or hypothesis generation for future studies, and this is not the primary aim of this study. Randomization is implemented to minimize the need for multivariate analyses.

In order to test a two sample non-inferiority hypothesis, a sample size of at least 46 in each arm will result in at least 80% power to conclude no more than 4% worse in SCC group vs. standard of care group (for continuous variables). Other test are only slightly less powered. Therefore, the investigators aim to enroll at least 46 patients in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Singletons born 35 0/7 to 36 6/7 weeks GA via vaginal delivery
* Vigorous - crying, good respiratory effort, good tone
* No major congenital malformation

Exclusion Criteria:

* Neonates born < 35 weeks GA
* Non-vigorous or needing resuscitation soon after birth
* Known major congenital malformation
* Maternal sedation or if clinically unstable per Labor & Delivery team

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Skin-to-skin interruptions | First hour of life
  The investigators will track the number of times skin-to-skin contact is disrupted within the first hour of life and document reasons for interruption.

SECONDARY OUTCOMES:
Risks for late-preterm neonates | Length of hospital stay
  The investigators will track the baby's temperature to monitor for hypothermia, glucose levels to monitor for hypoglycemia, and if there is transfer to the Neonatal Intensive Care Unit (NICU) anytime during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Bhola, MD, Principal Investigator — UH Cleveland Medical Center MacDonald Women's Hospital; Rebecca Walsh, MD, Principal Investigator — UH Cleveland Medical Center MacDonald Women's Hospital
Locations (1):
- UH Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT03585192/Prot_000.pdf